CLINICAL TRIAL: NCT02731209
Title: Functional Urodynamic Changes in Chronic Kidney Disease Patients and Does Insertion of Urinary Catheter in Chronic Kidney Disease Patients Grade 4 Delay the Need for Kidney Dialysis
Brief Title: Functional Urodynamic Changes in Chronic Kidney Disease Patients and Does Insertion of Urinary Catheter Delay the Need for Kidney Dialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf Harofeh MC (Other Government)
Responsible Party: Sponsor-Investigator, Assaf Harofeh MC, Medical doctor, Assaf-Harofeh Medical Center
Organization: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0308-15-ASF
Record Dates: First submitted 2016-02-22; First posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Urinary Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- catheter insertion for 2 weeks (Experimental): 50 randomized patients that will do urodynamic urinary examination and will be inserted urinary catheter for 2 weeks
  Interventions: Device: urinary catheter
- follow up (No Intervention): 50 randomized patients that will do urodynamic urinary examination and will be regularly followed by nephrologist

INTERVENTIONS:
Device: urinary catheter
  Arms: catheter insertion for 2 weeks

SUMMARY:
The aim of the investigators work is to describe the urodynamic results in the CKD (chronic kidney disease) grade 4 patients and to verify observations that urinary catheter may improve kidney function in those patients.

100 patients with CKD grade 4 will do urodynamic examination.

All patients will be randomized into two groups / the intervention group that will be inserted urinary catheter for 2 weeks and the follow up group. Kidney function will be monitored by creatinin values and the investigators will measure the time to dialysis in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* chronic kidney disease grade 4-5 (eGFR (estimated glomerular filtration rate) <30)
* eligible to sign a consent form

Exclusion Criteria:

* non controlled Diabetes Melitus (HbA1C>10%)
* not controlled HTN (Hypertension)
* cardiovascular event requiring cardiac stenting
* renal hydronephrosis or post void rest > 200CC according to US (Ultrasound)
* acute renal failure
* not eligible for urodynamics for any reason
* constant urinary catheter for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
kidney function change | At the time of urinary catheter insertion. Two weeks from the insertion and than after 8,16, 24, 32, 40 and 48 weeks after the urinary catheter insertion. (at total 52 weeks of follow up)
  measured by creatinine values mg/dL

SECONDARY OUTCOMES:
time to dialysis | at least 1 year from the time of catheter insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf ha Rofeh, MC, Zrifin, Israel